CLINICAL TRIAL: NCT03836170
Title: Analysis by High-throughput Sequencing: the Impact of Cholecystectomy on Gut Microbiome in Adults
Brief Title: Analysis of the Impact of Cholecystectomy on Gut Microbiome in Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: rjkls20190208
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: laparoscopic cholecystectomy; gut microbiota
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic cholecystectomy (Experimental): A laparoscopic cholecystectomy was performed to remove the gallbladder
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — A special catheter was inserted into the peritoneal cavity, and then about 2-5 liters of carbon dioxide was injected. After reaching a certain pressure, four small holes of 0.5-1.5cm were opened in the abdomen to dissect the structure of the triangle of the gallbladder. The gallbladder duct and gallbladder artery were cut off and closed, and then the entire gallbladder was removed.

SUMMARY:
Laparoscopic cholecystectomy (LC) is widely used in the gallbladder stone, gallbladder polyp, gallbladder cancer and other diseases. Some of the patients would develop diarrhea after surgery, and studies have reported an increased risk of colorectal cancer after LC. The aim of the present study was to examine the effects of LC on the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Gallbladder polyps diameter mm >10;
2. The history of the symptoms of patients with gallbladder stones, there was no history of acute attack in the past month;
3. Age <70 years old;
4. No serious systemic diseases such as diabetes, hypertension, heart disease, lung disease and so on/American anesthesia Association (ASA) grade I or II;
5. BMI<30;
6. Families have better care and observation, and away from the hospital within 1 hours; patients and their families understand the process of ambulatory surgery (24 hours) and the pros and cons.

Exclusion Criteria:

1. Less than 18 years old;
2. With previous gastric surgery ;
3. Major systemic diseases ;
4. Pregnancy or lactation;
5. The use of antibiotics or yogurt within 2 months before the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-05-20 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of gut microbiota after laparoscopic cholecystectomy | Three months and one year after completion of LC
  Three months and one year after completion of laparoscopic cholecystectomy therapy, gut microbiota was assessed by 16S rDNA high-throughput sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No